CLINICAL TRIAL: NCT01522872
Title: A Phase 1/2 Open-label Study to Assess the Safety, Tolerability and Preliminary Efficacy of TH-302, A Hypoxia-Activated Prodrug, and Dexamethasone With or Without Bortezomib or Pomalidomide in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Open-label Study of TH-302 and Dexamethasone With or Without Bortezomib or Pomalidomide in Subjects With Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-408
Record Dates: First submitted 2012-01-06; First posted 2012-02-01 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
Keywords: TH-302; Relapsed/Refractory Multiple Myeloma; Bortezomib; Phase 1/2; Hypoxia; Myeloma; Evofosfamide; Pomalidomide; Pimonidazole
MeSH Terms: conditions — Multiple Myeloma; Hypoxia; Neoplasms, Plasma Cell | interventions — TH 302; Dexamethasone; Bortezomib; pomalidomide

ARMS (4):
- Monotherapy TH-302 Dose Escalation (Experimental)
  Interventions: Drug: TH-302
- TH-302 and Dexamethasone Dose Expansion (Experimental)
  Interventions: Drug: TH-302 and Dexamethasone
- TH-302 Dose Escalation and Dexamethasone with Bortezomib (Experimental)
  Interventions: Drug: TH-302 Dose Escalation and Dexamethasone in Combination with Bortezomib
- TH-302 Dose Escalation and Dexamethasone with Pomalidomide (Experimental)
  Interventions: Drug: TH-302 Dose Escalation and Dexamethasone in Combination with Pomalidomide

INTERVENTIONS:
Drug: TH-302
  Arms: Monotherapy TH-302 Dose Escalation
Drug: TH-302 and Dexamethasone
  Arms: TH-302 and Dexamethasone Dose Expansion
Drug: TH-302 Dose Escalation and Dexamethasone in Combination with Bortezomib
  Arms: TH-302 Dose Escalation and Dexamethasone with Bortezomib
Drug: TH-302 Dose Escalation and Dexamethasone in Combination with Pomalidomide
  Arms: TH-302 Dose Escalation and Dexamethasone with Pomalidomide

SUMMARY:
This phase 2 study is designed to evaluate the safety and tolerability activity of TH-302 and dexamethasone with or without bortezomib or pomalidomide in subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is the initial study of TH-302 in subjects with relapsed/refractory multiple myeloma. It is an open-label dose-escalation study to determine the DLTs, MTD, safety and preliminary efficacy of TH-302 and dexamethasone with a Simon two-stage expansion at the MTD. The study will also investigate the DLTs, MTD, safety and preliminary efficacy of TH-302, dexamethasone and bortezomib; and the DLTs, MTD, safety and preliminary efficacy of TH-302, dexamethasone and pomalidomide. As such, the study is separated into four parts. Treatment will be administered until disease progression or unacceptable toxicity, or 12 cycles (Arm A, Arm B and Arm C) or 9 cycles (Arm D) have been completed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee.
3. Relapsed/refractory multiple myeloma for which no standard therapy options are anticipated to result in a durable remission.
4. Receipt of at least two prior therapies as indicated by protocol
5. Subjects with measurable disease
6. ECOG performance status of less than or equal to 2
7. Acceptable liver function
8. Acceptable renal function
9. Acceptable hematologic status
10. For Part A, B, C subjects: Women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception with their partner as indicated by protocol For Part D subjects: a negative serum pregnancy test is required within 10- 14 days prior to initiating with pomalidomide, AND a negative serum pregnancy test within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control at least 28 days before she starts taking pomalidomide.

    Women of childbearing potential must enroll into and follow all requirements of the POMALYST REMS program, which includes adhering to the scheduled pregnancy testing.

    Men must agree to use a latex or synthetic condom during sexual contact with women of child bearing potential even if they have had a vasectomy.

    All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure, or when a female patient misses her period or if there is any abnormality in her menstrual bleeding.
11. Subjects must adhere to the study visit schedule and other protocol requirements and receive outpatient therapy and laboratory monitoring at the institute that administers the study drug.

Exclusion Criteria

Subjects who meet any of the following exclusion criteria are not eligible to be enrolled in this study:

1. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes.)
2. Waldenstrom's macroglobulinemia
3. Localized radiation therapy to only measurable disease site(s) within 2 weeks of treatment
4. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, or unstable arrhythmia
5. Significant neuropathy (Grade 3 or 4, or Grade 2 with pain) at the time of enrollment or within 14 days before enrollment
6. Symptomatic brain metastases (unless previously treated and well controlled for a period of ≥ 3 months)
7. Severe chronic obstructive pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state leading to hypoxemia
8. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
9. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy within 14 days prior to the first dose
10. Previously treated malignancies, except for adequately treated non-melanoma skin cancer (basal cell or squamous cell), in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
11. Subjects who participated in an investigational drug or device study within 2 weeks prior to study entry
12. Known or suspected active infection with HIV, hepatitis A, hepatitis B, or hepatitis C
13. Subjects who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation similar to TH-302, bortezomib (for subjects enrolled in Part C only), pomalidomide (Part D), dexamethasone or pimonidazole
14. Females who are pregnant or breast-feeding
15. Concomitant psychiatric disease or medical condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
16. Unwillingness or inability to comply with the study protocol for any reason
17. Previous cytotoxic therapies for multiple myeloma within 3 weeks prior to study entry (2 weeks for biologic, novel therapy or corticosteroids)
18. Subjects who have been on hormone replacement less than 2 months (subjects on hormone replacement for at least 2 months will not be excluded provided the HRT regimen remains unchanged during the conduct of the study).
19. Prior peripheral stem cell transplant within 12 weeks of the start of study
20. Epilepsy or other convulsive disorder requiring active management
21. Prior therapy with a pomalidomide-containing regimen
22. Subjects on strong inducers or strong inhibitors of cytochrome P450 CYP3A4 or CYP1A2
23. Any other medical condition that in opinion of investigator would place patient at increased risk for toxicity during pomalidomide treatment (i.e. history of recurrent or serious thromboembolic events)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 30 days after last dose
Type of adverse events(AEs) | Up to 30 days after last dose
Severity of adverse events(AEs) | Up to 30 days after last dose
dose-limiting toxicities (DLTs) and the maximum tolerated dose (MTD) of TH-302 and dexamethasone with or without bortezomib or pomalidomide | 2 years
recommended Phase 2 dose for TH-302 and dexamethasone with or without bortezomib or pomalidomide | 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 12 weeks post treatment
Progression-free survival(PFS) | Up to 12 weeks post treatment
Duration of Response (DOR) | Up to 12 weeks post treatment
relationship between hypoxia within the bone marrow of subjects with relapsed/refractory multiple myeloma and response to TH-302 and dexamethasone with or without bortezomib or pomalidomide using markers of hypoxia | Up to 12 weeks post treatment
Maximum plasma concentration of TH-302 and bortezomib | Cycle 1 Day 1 predose and up to 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pacific Cancer Care, Monterey, California
  - Moffitt Cancer Center, Tampa, Florida
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The West Clinic, Southaven, Mississippi
  - New York Oncology Hematology, Albany, New York
  - New York Oncology Hematology, Hudson, New York
  - The West Clinic, Memphis, Tennessee